CLINICAL TRIAL: NCT07225504
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of Remibrutinib in Patients With Secondary Progressive Multiple Sclerosis
Brief Title: A Study to Evaluate the Efficacy and Safety of Remibrutinib in Secondary Progressive Multiple Sclerosis
Acronym: REMASTER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLOU064P12301; 2025-521546-23 (Other: EU Trial (CTIS) Number)
Expanded Access: NCT05170724 (Available)
Record Dates: First submitted 2025-11-04; First posted 2025-11-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Secondary Progressive Multiple Sclerosis (SPMS)
Keywords: MS; Multiple sclerosis; secondary progressive multiple sclerosis; SPMS; remibrutinib; LOU064; adult; Expanded Disability Status Scale; EDSS; McDonald diagnostic criteria
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — remibrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind on Core part and Open label on Extension part
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Remibrutinib (LOU064) (Experimental): Core Part: Remibrutinib film-coated tablet taken orally
  [Extension Part: Open-label remibrutinib film-coated tablet taken orally]
  Interventions: Drug: Remibrutinib (blinded); Drug: Remibrutinib (Open label)
- Placebo (Placebo Comparator): Core Part: Matching placebo film-coated tablet taken orally
  [Extension Part: Open-label remibrutinib film-coated tablet taken orally]
  Interventions: Drug: Placebo; Drug: Remibrutinib (Open label)

INTERVENTIONS:
Drug: Remibrutinib (blinded) — Remibrutinib (Blinded) active treatment, oral tablet
  Other Names: LOU064
  Arms: Remibrutinib (LOU064)
Drug: Placebo — Matching placebo (binded), oral tablet
  Arms: Placebo
Drug: Remibrutinib (Open label) — Remibrutinib (Open Label), oral tablet
  Other Names: LOU064

SUMMARY:
The purpose of this study is to provide efficacy and safety data for remibrutinib in patients with secondary progressive multiple sclerosis (SPMS)

DETAILED DESCRIPTION:
This is a Phase III, randomized, double-blind, placebo-controlled, multi-center, parallel-group, event-driven study to evaluate the efficacy, safety and tolerability of remibrutinib in SPMS patients. Approximately 1275 eligible participants will be randomized to receive either remibrutinib or matching placebo.

The study consists of an event-driven Core Part with double-blind treatment, followed by an Extension Part with open-label remibrutinib treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to any assessment performed.
* Male or female participants aged 18-65 (inclusive) at Screening.
* Diagnosis of SPMS according to the 2017 revised McDonald criteria (Thompson et al 2018) at Screening.
* Absence of documented clinical relapses in the 24 months before Screening and randomization.
* EDSS score of 3.0 to 6.0 (inclusive) at Screening.
* Documented evidence of disability progression in the 12 months before Screening.

Exclusion Criteria:

* Unwilling or unable to undergo MRI scans as per protocol (for example, claustrophobia, or presents absolute contraindications to MRI (e.g., metallic implants, metallic foreign bodies, pacemaker, defibrillator)).
* History of clinically significant central nervous system (CNS) disease (e.g. stroke, traumatic brain or spinal injury, history or presence of myelopathy) or neurological disorders which may mimic multiple sclerosis (MS).
* Ongoing substance abuse (drug or alcohol) or any other factor (e.g. serious psychiatric condition) that may interfere with the participant's ability to cooperate and comply with the study procedures.
* Participants with history of confirmed Progressive Multifocal Leukoencephalopathy (PML) or neurological symptoms consistent with PML.
* Women of childbearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant from menarche until becoming post-menopausal, unless they are using highly effective methods of contraception (failure rate < 1% per year) while taking study treatment and for at least 1 week after stopping study treatment.
* Significant bleeding risk or coagulation disorders, at Screening.
* Use of exclusionary medication prior to Screening/randomization as listed in the protocol.

Other protocol-defined inclusion/exclusion critria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1275 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2030-12-03 (Estimated); Study Completion 2034-01-02 (Estimated)

PRIMARY OUTCOMES:
Time to 6-month confirmed disability progression (6mCDP) on Expanded Disability Status Scale (EDSS) | From baseline up to approximately 5 years
  The EDSS is an ordinal scale used for assessing neurologic impairment in MS based on a neurological examination. It consists of scores in each of seven functional systems and an ambulation score that are then combined to determine the EDSS steps (ranging from 0 (normal) to 10 (death due to MS)).
  6mCDP is defined as an increase from baseline in EDSS sustained for at least 6 months.

SECONDARY OUTCOMES:
Time to 3-month confirmed disability progression (3mCDP) on EDSS | From baseline up to approximately 5 years
  The EDSS is an ordinal scale used for assessing neurologic impairment in MS based on a neurological examination. It consists of scores in each of seven functional systems and an ambulation score that are then combined to determine the EDSS steps (ranging from 0 (normal) to 10 (death due to MS)).
  3mCDP is defined as an increase from baseline in EDSS sustained for at least 3 months.
Time to 6-month confirmed disability improvement (6mCDI) on EDSS | From baseline up to approximately 5 years
  The EDSS is an ordinal scale used for assessing neurologic impairment in MS based on a neurological examination. It consists of scores in each of seven functional systems and an ambulation score that are then combined to determine the EDSS steps (ranging from 0 (normal) to 10 (death due to MS)).
  A 6mCDI is defined as a decrease from baseline in EDSS sustained for at least 6 months.
Time to 3-month worsening by at least 20% in Timed 25-Foot Walk (T25FW) | From baseline up to approximately 5 years
  The T25FW is an ambulation measurement assessing speed of walking: a timed (in seconds) walk of 25 feet (7.62 meters). Longer time indicates poorer lower limb function.
  3-month worsening by at least 20% in T25FW is defined as an increase from baseline in T25FW of at least 20% sustained for at least 3 months.
Time to 3-month worsening by at least 20% in 9-Hole Peg Test (9-HPT) | From baseline up to approximately 5 years
  The 9-HPT is an objective quantitative test of neurological function. It is measured to assess both right and left arm scores, the metric is the time, in seconds, required to insert and remove 9 pegs. Longer time indicates poorer upper limb function.
  A 3-month worsening by at least 20% in 9-HPT is defined as an increase from baseline in 9-HPT of at least 20% sustained for at least 3 months
Annualized rate of new or enlarging T2 lesions | From baseline up to approximately 5 years
  Number of new or enlarging T2 lesions per year based on MRI
Annualized rate of brain atrophy | From baseline up to approximately 5 years
  Percentage change in brain volume relative to baseline per year based on MRI assessments
Time to 6-month worsening by at least 4 points in Symbol Digit Modalities Test (SDMT) | From baseline up to approximately 5 years
  The SDMT is a sensitive and specific test to assess information processing speed which is typically affected in cognitively impaired MS participants, The test scoring is calculated based on the number of correct answers in 90 seconds.
  A 6-month worsening by at least 4 points in SDMT is defined as an increase from baseline in SDMT of at least 4 points sustained for at least 6 months.
Number of participants with Adverse events and Serious adverse events (SAE) | From baseline up to approximately 5 years
  Incidence of adverse events including changes in laboratory data, vital signs, electrocardiogram (ECG) and Columbia Suicide Severity Rating Scale (C-SSRS) qualifying and reported as AEs.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (8):
  - Alabama Neurology Associates PC, Birmingham, Alabama
  - AZ Integrated Neuro and Spine, Phoenix, Arizona
  - Neurology of Central FL Res Ctr, Altamonte Springs, Florida
  - Orlando Health Clinical Trials, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Mid Atlantic Epilepsy and Sleep Ctr, Bethesda, Maryland
  - Michigan Institute of Neurological, Farmington Hills, Michigan
  - Neurology Clinic PC, Cordova, Tennessee
- Australia (2):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Heidelberg, Victoria
- Canada (2):
  - Novartis Investigative Site, Lévis, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- Israel (5):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
  - Novartis Investigative Site, Ẕerifin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com